CLINICAL TRIAL: NCT01356004
Title: Live Attenuated Varicella Vaccine: A New Effective Adjuvant Weapon in the Battlefield Against Severe Resistant Psoriasis, a Randomized Controlled Trial
Brief Title: Effective Study of Live Attenuated Varicella Vaccine to Treat Severe Resistant Psoriasis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Prof. Mohammad El Darouti, Faculty of Medicine, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CairoU
Record Dates: First submitted 2011-05-17; First posted 2011-05-19 (Estimated); Last update posted 2011-05-19 (Estimated); Status verified 2011-01

CONDITIONS: Psoriasis
Keywords: severe resistant
MeSH Terms: conditions — Psoriasis | interventions — Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- chicken pox vaccine, efficacy (Experimental)
  Interventions: Drug: live attenuated chicken pox vaccine
- saline, efficacy (Placebo Comparator)
  Interventions: Drug: saline, efficacy

INTERVENTIONS:
Drug: live attenuated chicken pox vaccine — Each immunizing dose was given subcutaneously (SC) in the form of 0.5 ml reconstituted vaccine which contains not less than 1033 plaque forming units (PFU) of the attenuated varicella-zoster-virus (VZV), which meets the World Health Organization (WHO) requirements for biological substances and for varicella vaccines. Doses were given 3 weeks apart for a total duration of 12 weeks (3 months).
  Arms: chicken pox vaccine, efficacy
Drug: saline, efficacy — 4 doses of SC saline (0.5 ml) -as a placebo- in the same pattern as group A patients
  Arms: saline, efficacy

SUMMARY:
Immunotherapy was reported in the treatment of psoriasis. Treatment of resistant psoriasis may be difficult and cyclosporine can induce some remission.

The investigators hypothesized that the combined use of live attenuated varicella vaccine as an adjuvant therapy to low dose cyclosporine in the treatment of severe resistant psoriasis can give positive responses.

ELIGIBILITY:
Inclusion Criteria:

* Severe psoriasis: At least 30% of body involved) according to the rule of nine.
* Resistance to conventional therapy (PUVA, methotrexate, retinoids):

(Maximum PASI 50% improvement while on treatment for a duration not less than 6 months).

* Immunologically competent individuals with
* Seropositive for the varicella antibodies

Exclusion Criteria:

* Any contraindication to live attenuated varicella vaccine
* Any contraindication to cyclosporine

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2010-01; Primary Completion 2010-05 (Actual); Study Completion 2010-11 (Actual)

PRIMARY OUTCOMES:
Number of Participants with PASI score improvement as a Measure of effective treatment | 12 weeks
  the clinical evaluation of our patients through the Psoriasis Area Severity Index (PASI) score calculation at each visit.
  The final patient's response was rated according to the physician global assessment (PGA) based on the final improvement of the PASI score as worse, poor (0-24% improvement in PASI), fair (25-50% improvement in PASI), good (50-74% improvement in PASI), excellent (75-99% improvement in PASI), or cleared (100% improvement in PASI).

SECONDARY OUTCOMES:
Number of Participants with Adverse Events as a Measure of Safety and Tolerability | 12 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Cairo, Egypt